CLINICAL TRIAL: NCT06130280
Title: Ablative Dose Single Fraction MRguided Colorectal Liver Metastasis SBRT
Brief Title: A Study of Single Fraction Stereotactic Body Radiation Therapy (SBRT) Guided by Magnetic Resonance Imaging (MRI) in People With Liver Metastasis From Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-285
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Single Fraction Stereotactic Body Radiation Therapy (SBRT); Magnetic Resonance Imaging (MRI); 23-285
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A phase II prospective trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR Guided Single Fraction Stereotactic Body Radiation Therapy (SBRT) (Experimental): Participants will undergo simulation including Gd-EOB-DTPAenhanced MR and planning using minimal margins. Ten days later (+/- 3 days) participants will receive 40Gy single fraction treatment on Elekta Unity using Gd-EOB-DTPA-enhanced MR for image guidance and on-line adaptive replanning.
  Interventions: Radiation: MR Guided Single Fraction Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: MR Guided Single Fraction Stereotactic Body Radiation Therapy (SBRT) — 40Gy single fraction treatment on Elekta Unity using Gd-EOB-DTPA-enhanced MR for image guidance.

SUMMARY:
The researchers are doing this study to see if one session of high-dose contrast-enhanced MRI-guided SBRT (stereotactic body radiation therapy) is effective for colorectal cancer that has spread to the liver. The researchers will evaluate how well the study treatment can prevent the liver metastasis from growing and spreading. In addition, they will see whether it causes any side effects and whether there are any characteristics of the research MRI images that can predict response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Histologically confirmed colorectal carcinoma and evidence of liver metastasis on imaging
* ECOG 0-2
* <=3 liver lesions measurable on contrast enhanced diagnostic MRI with combined size (sum of longest diameters) < 7 cm, and individual size < 5cm. (Subsequent simulation scans will not be used for eligibility assessment. In case of significant change in size exceeding 1cm, the individual participants can continue on the protocol provided all normal tissue contraints are met during planning).
* Lesion location at least ≥ 2 cm of main, right and left portal vein on the baseline diagnostic MRI. (Subsequent simulation scans will not be used for eligibility assessment. In case of significant change in the distance between the lesion edge and critical structure exceeding 1cm, the individual participants can continue on the protocol provided all normal tissue contraints are met during planning ).
* Lesion location at least ≥ 1.5 cm of luminal gastrointestinal tract (stomach, small and large bowel). (Subsequent simulation scans will not be used for eligibility assessment. In case of significant change in the distance between the lesion edge and critical structure exceeding 1cm, the individual participants can continue on the protocol provided all normal tissue contraints are met during planning).
* Lesion location ≥ 0.5 cm of diaphragm
* Preserved liver function as defined by:

  * Albumin > 2 g/dl
  * < AST/ ALT ≤ 5 x ULN
  * Total Bilirubin ≤ 1.5 x UL
* Negative serum pregnancy test within 14 days prior to simulation and MRgRT for women of childbearing potential
* Any prior systemic or hepatic artery intraarterial pump (HAIP) chemotherapy is permitted with a washout of 2 weeks
* Any prior treatment with FDA-approved or investigational biologics or novel molecularly targeted therapies, including oral or IV formulations, are permitted with a washout of 1 weeks or 4 half-lives, which ever is longer
* Extrahepatic disease outside the liver is permitted
* Prior liver resection is permitted provided there is enough liver parenchyma to meet normal tissue contraints
* Prior liver-directed RT is permitted provided departmental normal tissue constraints for re-irradiation can be met
* Review by HBP DMT prior to enrollment

Exclusion Criteria:

* Any history of cirrhosis
* History of hepatic radioembolization or selective internal radiation therapy (SIRT)
* History of inflammatory bowel disease that precludes liver RT (at the discretion of the treating radiation oncologist).
* Current pregnancy or breastfeeding
* Men or women not using effective contraception.
* Contraindication to or inability to undergo an MR scan, including, but not limited to the history of MR unsafe implants, any implanted cardiac pacemakers or deffibrilators, history of claustrophobia, and contraindications to Gd-EOB-DTPA contrast agent.
* Concurrent anti-neoplastic therapy of any kind defined as receipt within 1 week of RT administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Local control rate CRC liver metastasis | 1 year
  by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Reyngold, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm